CLINICAL TRIAL: NCT02679547
Title: The Effect of Breastfeeding on the Development of Appendicitis in Adults
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Collaborators: Istanbul Training and Research Hospital (Other Government); Bezmialem Vakif University (Other); Arnavutkoy State Hospital (Other); Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ufuk Oguz Idiz, M.D, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: Breastfeeding
Record Dates: First submitted 2016-02-03; First posted 2016-02-10 (Estimated); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Appendicitis
Keywords: Appendix; Breastfeeding; Adult
MeSH Terms: conditions — Appendicitis; Breast Feeding | interventions — Lactation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Appendicitis: The patients with appendicitis
  Interventions: Other: Breastfeeding
- Control: The participants without appendicitis
  Interventions: Other: Breastfeeding

INTERVENTIONS:
Other: Breastfeeding — All of the participants and patients will have a questionnaire about their breastfeeding

SUMMARY:
Appendectomy is the most common emergent operative procedure performed worldwide. In this study investigators will investigate if there is a relationship between breast feeding and appendicitis in adults.

DETAILED DESCRIPTION:
Acute appendicitis accounts for the commonest indication for emergency visits during daily surgical practice. Breast feeding is very important both mother and the child. For the infant, breast feeding has an important role on the maturity of immune system. In the literature search, there are a little studies about the relationship between the breast feeding and appendicitis. In the literature, some studies suggests that the breast feeding may possibly give protection against the development of appendicitis. But the number of the patients and the control groups are limited. Because of that the investigators have planned to make this study with a lot of number of patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects has pathologically proven appendicitis for appendicitis group.

Exclusion Criteria:

* Subjects has American Society of Anesthesiologists Physical Status classification 4,
* Subject has pregnancy,
* Subject has malignity,
* Subject has chronic illness,
* Subjects who won't accept to join the study
* Subjects who don't have family members

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 500 patients who has pathologically proven appendicitis, and 1000 participants without appendicitis.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2016-01; Primary Completion 2019-12 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
The breastfeeding status questionnaire in the appendicitis patients and participants without appendicitis | 2 days
  500 patients who have pathologically proven appendicitis and 1000 controls without appendicitis will be asked the question which is "How long did you had breast feeding?". The patients and the participants will be in the same age groups. Also the same question will be asked to at least one of the family member (mother, father, older brother or older sister). The breastfeeding status will be in three group ( 0-2 months, 2-6 months and >6 months)

CONTACTS AND LOCATIONS:
Locations (5):
- Turkey (Türkiye) (5):
  - Bursa Yuksek Ihtisas Training and Research Hospital, Bursa
  - Sisli Etfal Training and Research Hospital, Istanbul
  - Arnavutkoy State Hospital, Istanbul
  - Bezmialem Vakif University, Istanbul
  - Istanbul Training and Research Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided
Because the time period of this study is very short

REFERENCES:
- [Background] Minniti F, Comberiati P, Munblit D, Piacentini GL, Antoniazzi E, Zanoni L, Boner AL, Peroni DG. Breast-milk characteristics protecting against allergy. Endocr Metab Immune Disord Drug Targets. 2014 Mar;14(1):9-15. doi: 10.2174/1871530314666140121145045. PMID 24450452
- [Background] Pisacane A, de Luca U, Impagliazzo N, Russo M, De Caprio C, Caracciolo G. Breast feeding and acute appendicitis. BMJ. 1995 Apr 1;310(6983):836-7. doi: 10.1136/bmj.310.6983.836. No abstract available. PMID 7711621
- [Background] Alves JG, Figueiroa JN, Barros I. Does breast feeding provide protection against acute appendicitis? A case-control study. Trop Doct. 2008 Oct;38(4):235-6. doi: 10.1258/td.2008.070404. PMID 18820196